CLINICAL TRIAL: NCT05841498
Title: A Single-blinded Sham-controlled Crossover Trial to Evaluate the Effect of Immunoadsorption on Post-Corona Virus Disease (COVID)-Syndrome
Brief Title: Immunoadsorption Study Mainz in Adults With Post-COVID Syndrome
Acronym: IAMPOCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Mainz (Other)
Responsible Party: Principal Investigator, Prof. Dr. Julia Weinmann-Menke, Univ. Prof. Dr. med., University Medical Center Mainz
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IAMPOCO
Record Dates: First submitted 2023-04-25; First posted 2023-05-03 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Post-COVID-19 Syndrome; Post-COVID Syndrome; Post COVID-19 Condition
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Plasmapheresis

STUDY DESIGN:
Intervention Model Description: Single-blinded, randomized, sham-controlled, crossover trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immunoadsorption (Active Comparator): Immunoadsorption will be conducted with the Plasauto Sigma extracorporeal therapy system in combination with the TR-350 adsorber (Addendum February 2024: or with the Miltenyi Life-21 system in combination with the Ig-Omni adsorber) over 7 days (3 times daily, 2 times every other day). During each session 2-2.5 times the participant's plasma volume will be treated. This therapy regimen is proven by studies with groups of patients suffering from other autoimmune diseases (Boedecker, Luessi et al. 2022). The material needed for the immunoadsorption is provided by Diamed, the provider of Plasauto Sigma and TR-350 adsorber (Addendum February 2024: or by Miltenyi Biotec, the Provider of Life-21 and IgOmni) . To exclude possible beneficial or adverse effects of heparin on participants' symptoms, regional anticoagulation will be performed using citrate.
  This is a cross-over study: Each participant will receive immunoadsorption and sham treatment with a wash-out period of 8 weeks in between.
  Interventions: Device: Immunoadsorption
- Sham-apheresis (Sham Comparator): The sham procedure will also be conducted with the Plasauto Sigma extracorporeal therapy system (Addendum February 2024: or the Miltenyi Life-21 therapy system) without an inserted adsorber. To ensure that sham treatment is indistinguishable from immunoadsorption for the subjects, the therapy regimen is identical except for the missing adsorber. For both verum therapy and sham procedure, the devices are placed behind a portable wall and covered with a curtain not visible to the patient. However, since the setup of the machines differs depending on the procedure, it is not possible to blind the supervising staff as well. To exclude possible beneficial or adverse effects of heparin on participants' symptoms, regional anticoagulation will be performed using citrate. If a subject does not have sufficiently large peripheral veins, a large-bore central venous catheter will be placed for both IA and sham treatments.
  Interventions: Device: Sham-apheresis

INTERVENTIONS:
Device: Immunoadsorption — Immunoadsorption (IA) is a well-established extracorporeal therapy for several autoimmune diseases such as systemic lupus. Its therapeutic effect is based on the removal of antibodies (ABs) from the plasma including auto-ABs and it is used if an immediate response to therapy is necessary. Side effects (SE) of the IA are rare, but angiotensin-converting enzyme (ACE)-inhibitors are prohibited concomitant medication. Notable SE may include increased susceptibility to infection, transient disorders of blood coagulation, or allergic reactions to materials of the adsorber or tubing system. To ensure an effective therapy, a blood flow of at least 45 ml/min is necessary. In some patients, adequate blood flow can be achieved by cannulation of peripheral veins but in most patients is the placement of a central venous catheter necessary. Central venous catheter placement carries potential risks such as injury to the lung or mispuncture of the carotid artery.
  Arms: Immunoadsorption
Device: Sham-apheresis — Sham-apheresis is a procedure without any known therapeutic effects. As there are no known therapeutic effects there are also no known side effects excepted the risk of an allergic reaction to materials of the tubing system or to citrate, which is necessary to prevent clotting inside the extracorporeal system. To ensure a smooth operation a blood-flow of at least 45ml/min is necessary. In some patients, adequate blood flow can be achieved by cannulation of peripheral veins. However, in most patients, placement of a Shaldon catheter into the internal jugular vein is necessary. Shaldon catheter placement carries other potential risks such as injury to the lung resulting in pneumothorax or mispuncture of the carotid artery. However, since the catheter placement is sonography-guided, the risks for such adverse events are minimized.
  Arms: Sham-apheresis

SUMMARY:
The aim of this study is to evaluate the efficiency and safety of immunoadsorption for the treatment of post-COVID syndrome (PCS).

Efficacy will be measured (1) subjectively as an improvement of the score of questionnaires like the multidimensional fatigue inventory (MFI-20), Chalder fatigue scale, Bell-score, modified medical research council dyspnea scale (mMRC) and the Post-COVID functional scale (PCFS) and (2) objectively as an improvement in neurocognitive testing with the Montreal cognitive assessment (MoCA) and the improvement of the hand-grip strength.

40 participants with symptoms of PCS and a PCFS score of at least 2 will be included in each group (Addendum from February 2024: An additional 40 patients with the same inclusion and exclusion criteria will be treated using the devices and materials of another manufacturer, following the same design, and the results will be evaluated separately.). After excluding other causes of the symptoms and evaluating the baseline burden of symptoms, each participant will undergo 5 sessions of immunoadsorption with an immunoglobulin-binding adsorber and 5 sham treatments, or vice versa. The order of treatments (immunoadsorption first or sham first) will be randomized. Each participant will be blinded to the type of treatment they receive. An 8-week therapy-free period will separate the two treatment blocks. All examinations will be conducted before the first treatment, 2 weeks after the first treatment cycle, before the second treatment cycle, and 2 and 6 weeks after the second treatment cycle.

The results of the study will inform future treatment strategies for PCS and will contribute to a better understanding of the pathophysiological insights behind the ongoing symptoms.

DETAILED DESCRIPTION:
Post-COVID syndrome (PCS) refers to symptoms that develop 3 months from the onset of COVID-19 with symptoms that last for at least 2 months and cannot be explained by an alternative diagnosis (Soriano, Murthy et al. 2022). The nature of the symptoms has not been a factor in the definition of PCS. The prevalence of PCS is estimated to be 43% of all severe acute respiratory syndrom coronavirus 2 (SARS-COV-2)-infected patients, with hospitalized patients more likely to suffer from persistent symptoms (54%) than non-hospitalized patients (32%). Women are more likely to experience PCS than men (incidence, 49% vs 32%, respectively) (Chen, Haupert et al. 2022). The most common symptoms are fatigue (23%), memory impairment (14%), dyspnea (13%), sleep disturbances (11%), and joint pain (10%) (Chen, Haupert et al. 2022). Headaches, myalgia, anxiety or depression are also frequently reported.

In terms of the type, variety and duration of symptoms, PCS resembles a clinical picture observed after various viral infections, such as Eppstein-Barr virus, herpes simplex virus or influenza virus, namely myalgic encephalomyelitis and chronic fatigue syndrome (ME/CFS). Here, too, patients mainly suffer from fatigue, impaired concentration and memory, and non-restorative sleep. Some authors consider post-COVID as a form of ME/CFS triggered by the SARS-CoV-2 infection or the immune response to the infection. The underlying pathophysiology likely depends on the different viruses but is incompletely understood. Similarly, the causes of PCS are unclear to date. Autoimmunity is suspected to play a major role in all post-virus syndromes. It may be triggered by the defense against infections and is probably maintained by similarity of endogenous proteins with pathogen components (molecular mimicry). In the context of this autoimmunity, antibodies against endogenous structures can also be formed, such as antinuclear antibodies, which are directed against components of the cell nuclei. Antibodies against α- and β-adrenergic receptors and muscarinic acetylcholine receptors, among others, have been detected in patients suffering from ME/CFS as well as in patients with PCS.

Many patients are limited in their daily lives by the symptoms that develop or persist after SARS-COV-2-infection and suffer from a diminished quality of life. To date, there is little evidence on potential therapies for these complaints. Immunoadsorption (IA) efficiently removes (auto-)antibodies from the circulation and has been proposed as a potential therapy for PCS. The current trial will investigate the efficacy of IA for the treatment of PCS.

40 participants with PCS and a PCFS-score of at least 2 will be included in each. Each participant will undergo 5 sessions of IA with an immunoglobulin-binding adsorber and 5 sham treatments or vice versa. Sham treatment will be performed in the same ways as IA, but the IA device will not be set up with an adsorber. The order of treatments (immunoadsorption first or sham first) will be randomized. The participants are blinded to the order of treatments. An intervention-free interval of 8 weeks will separate both treatment blocks (Addendum from February 2024: 40 patients additional with the same inclusion and exclusion criteria will be treated using the devices and materials of another manufacturer, following the same design, and the results will be evaluated separately.).

The primary outcome of the study is the efficacy of IA vs. sham, measured as changes in the PCFS (0-4), Chalder-fatigue scale (0-33), MFI-20 (20-100), Bell score (0-100), montreal cognitive assesment and the hand-grip strength before therapy compared to values after immunoadsorption and after sham-treatment. Secondary outcomes are (1) the number and severity of adverse events, (2) the prevalence of auto-antibodies like antinuclear antibodies, antibodies against adrenoreceptors and antibodies against muscarinic acetylcholine receptors in patients with PCS and (3) the change in concentration of the auto-antibodies in context of therapy and sham-treatment. In addition, various assessments (Complete blood count with differential, Antinuclear antibody Thyroid-stimulating hormone, C-reactive protein, Vitamin B12, Vitamin D, 25-dihydroxy, Ferritin, Urinalysis, ECG, spirometry, psychological questionaires) will be performed during screening period to be able to exclude other diseases as the cause of the PCS symptoms. In addition, safety-relevant parameters such as heart rate, blood pressure, electrolyte concentra-tions, fibrinogen concentration and the concentration of the immunoglobulin fractions are measured before and after each treatment.

The results of the study will inform future treatment strategies for PCS and will contribute to a better understanding of the pathophysiological insights behind the ongoing symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Meeting the WHO diagnostic criteria for PCS
* Written informed consent to participate in the study
* Previous participation in the Gutenberg Post-Covid Study or previously conducted comparable preliminary examinations
* Minimum age of 18 years
* Value on the Post-COVID functional scale of at least 2

Exclusion Criteria:

* Psychiatric diagnosis
* Allergy to adsorber materials, materials of the tubing systems or to the substances used for immunoadsorption
* Pregnancy
* Medical contraindications to immunoadsorption such as severe blood clotting disorders or immunodeficiency syndromes
* Existing antibody-mediated autoimmune disease
* Intake of ACE-inhibitors 7 days prior to the inclusion in to the study or during the study period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-05-08 (Actual); Primary Completion 2025-05-12 (Actual); Study Completion 2025-05-12 (Actual)

PRIMARY OUTCOMES:
Improvement of Post-COVID symptoms as measured by PCFS score | 2 weeks after completion of immunoadsorption and sham-apheresis
  The PCFS serves as a self-report instrument to better objectify perceived symptom severity at Post-COVID. Patients are asked to describe states presented as a questionnaire. A value is assigned to each described state. The greater the symptom severity is described by the condition, the greater the score from 0-4. The PCFS has been validated in cohorts of patients with Post-COVID-syndrome and is therefore particularly suitable for assessing symptom severity.
Change of physical and/or mental fatigue as measured by Chalder-Fatigue-scale | 2 weeks after completion of immunoadsorption and sham-apheresis
  The Chalder Fatigue Scale is an 11-item question battery that captures two dimensions of fatigue symptomatology, both the assessment of physical functioning and the assessment of mental functioning. Each question is answered using a 4-point Likert scale. The answering takes an average of 2-3 minutes and a re-survey can be done every 4 weeks.
Change of impairment due to fatigue as measured by Bell-Score | 2 weeks after completion of immunoadsorption and sham-apheresis
  The Bell score is an assessment instrument that can be collected by both the patient and the examiner and measures the degree of restriction in daily life caused by fatigue symptoms. In 11 grades, the restriction can be indicated from 0 (bedridden) to 100 (no restrictions, normal resilience in all activities of daily living).
Change of physical and/or mental fatigue as measured by MFI-20 | 2 weeks after completion of immunoadsorption and sham-apheresis
  The MFI-20 captures the phenomenon of fatigue in the 5 subscales general fatigue, physical fatigue, reduced activity, reduced motivation, and mental fatigue. It is a self-report questionnaire in which patients rate statements such as "I was able to concentrate well" or "I was rested" in 5 levels for the latter time, including today. The result is a score in the range from 20-100 whereby a higher score indicates more severe fatigue.
Change of Hand grip strength measured as hand-grip-strength test with a dynamometer | 2 weeks after completion of immunoadsorption and sham-apheresis
  Grip strength serves as a surrogate parameter for physical performance or changes in it. Grip strength is measured three times on each hand in neutral position using a dynamometer and the mean value is documented.
Change of cognitive impairment as measured by Montreal cognitive assesment (MoCA) | 2 weeks after completion of immunoadsorption and sham-apheresis
  The Montreal Cognitive Assessment (MocA) is used to test various neurocognitive functions. It is a ten-minute test with various tasks that can be scored with a total of up to 30 points. It tests abilities in the areas of memory, attention, verbal abstraction, visuospatial abilities, concentration and language comprehension.

SECONDARY OUTCOMES:
number of treatment-emergent adverse events (TEAE), serious adverse events and discontinuation of therapy because of adverse events | 2 weeks after completion of immunoadsorption and sham-apheresis
  1. The number of treatment-emergent adverse events (TEAE), serious adverse events and discontinuation of therapy because of adverse events and the comparison of them under immunoadsorption with the number of events under sham apheresis. Events are recorded for comparison two weeks after the end of each treatment cycle.
Prevalence of anti-adrenergic and anti-muscarinic autoantibodies in patients with PCS: | at the time of the first examination before randomization for the first treatment-modality
  1. Proportion of subjects with evidence of anti-α1-adrenoreceptor antibodies (AB)
  2. Proportion of subjects with evidence of anti-α2-adrenoreceptor AB
  3. Proportion of subjects with evidence of anti-β1-adrenoreceptor-AB
  4. Proportion of subjects with evidence of anti-β2-adrenoreceptor AB
  5. Proportion of subjects with evidence of anti-β3-adrenoreceptor-AB
  6. Proportion of subjects with detection of anti- M1 acetylcholine receptor AB
  7. Proportion of subjects with detection of anti-M2 acetylcholine receptor AB
  8. Proportion of subjects with detection of anti-M3 acetylcholine receptor-AB
  9. Proportion of subjects with detection of anti-M4 acetylcholine receptor-AB
3. Concentration of autoantibodies before and after IA and sham treatment (before therapy cycle 1/after therapy cycle1 as well as before therapy cycle 2/after therapy cycle 2) | before therapy cycle 1/after therapy cycle1 as well as before therapy cycle 2/after therapy cycle 2
  1. Concentration anti-α1-adrenoreceptor antibodies (AB)
  2. Concentration of anti-α2-adrenoreceptor AB
  3. Concentration of anti-β1-adrenoreceptor-AB
  4. Concentration of anti-β2-adrenoreceptor AB
  5. Concentration of anti-β3-adrenoreceptor-AB
  6. Concentration of anti- M1 acetylcholine receptor AB
  7. Concentration of anti-M2 acetylcholine receptor AB
  8. Concentration of anti-M3 acetylcholine receptor-AB
  9. Concentration of anti-M4 acetylcholine receptor-AB

CONTACTS AND LOCATIONS:
Locations (1):
- UNIVERSITÄTSMEDIZIN der Johannes Gutenberg-Universität Mainz I. Medizinische Klinik und Poliklinik, Mainz, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bateman L, Bested AC, Bonilla HF, Chheda BV, Chu L, Curtin JM, Dempsey TT, Dimmock ME, Dowell TG, Felsenstein D, Kaufman DL, Klimas NG, Komaroff AL, Lapp CW, Levine SM, Montoya JG, Natelson BH, Peterson DL, Podell RN, Rey IR, Ruhoy IS, Vera-Nunez MA, Yellman BP. Myalgic Encephalomyelitis/Chronic Fatigue Syndrome: Essentials of Diagnosis and Management. Mayo Clin Proc. 2021 Nov;96(11):2861-2878. doi: 10.1016/j.mayocp.2021.07.004. Epub 2021 Aug 25. PMID 34454716
- [Background] Boedecker SC, Luessi F, Engel S, Kraus D, Klimpke P, Holtz S, Meinek M, Marczynski P, Weinmann A, Weinmann-Menke J. Immunoadsorption and plasma exchange-Efficient treatment options for neurological autoimmune diseases. J Clin Apher. 2022 Feb;37(1):70-81. doi: 10.1002/jca.21953. Epub 2021 Dec 14. PMID 34904748
- [Background] Chen C, Haupert SR, Zimmermann L, Shi X, Fritsche LG, Mukherjee B. Global Prevalence of Post-Coronavirus Disease 2019 (COVID-19) Condition or Long COVID: A Meta-Analysis and Systematic Review. J Infect Dis. 2022 Nov 1;226(9):1593-1607. doi: 10.1093/infdis/jiac136. PMID 35429399
- [Background] Poenaru S, Abdallah SJ, Corrales-Medina V, Cowan J. COVID-19 and post-infectious myalgic encephalomyelitis/chronic fatigue syndrome: a narrative review. Ther Adv Infect Dis. 2021 Apr 20;8:20499361211009385. doi: 10.1177/20499361211009385. eCollection 2021 Jan-Dec. PMID 33959278
- [Background] Son K, Jamil R, Chowdhury A, Mukherjee M, Venegas C, Miyasaki K, Zhang K, Patel Z, Salter B, Yuen ACY, Lau KS, Cowbrough B, Radford K, Huang C, Kjarsgaard M, Dvorkin-Gheva A, Smith J, Li QZ, Waserman S, Ryerson CJ, Nair P, Ho T, Balakrishnan N, Nazy I, Bowdish DME, Svenningsen S, Carlsten C, Mukherjee M. Circulating anti-nuclear autoantibodies in COVID-19 survivors predict long COVID symptoms. Eur Respir J. 2023 Jan 12;61(1):2200970. doi: 10.1183/13993003.00970-2022. Print 2023 Jan. PMID 36137590
- [Background] Soriano JB, Murthy S, Marshall JC, Relan P, Diaz JV; WHO Clinical Case Definition Working Group on Post-COVID-19 Condition. A clinical case definition of post-COVID-19 condition by a Delphi consensus. Lancet Infect Dis. 2022 Apr;22(4):e102-e107. doi: 10.1016/S1473-3099(21)00703-9. Epub 2021 Dec 21. PMID 34951953
- [Background] Sotzny F, Filgueiras IS, Kedor C, Freitag H, Wittke K, Bauer S, Sepulveda N, Mathias da Fonseca DL, Baiocchi GC, Marques AHC, Kim M, Lange T, Placa DR, Luebber F, Paulus FM, De Vito R, Jurisica I, Schulze-Forster K, Paul F, Bellmann-Strobl J, Rust R, Hoppmann U, Shoenfeld Y, Riemekasten G, Heidecke H, Cabral-Marques O, Scheibenbogen C. Dysregulated autoantibodies targeting vaso- and immunoregulatory receptors in Post COVID Syndrome correlate with symptom severity. Front Immunol. 2022 Sep 27;13:981532. doi: 10.3389/fimmu.2022.981532. eCollection 2022. PMID 36238301
- [Derived] Stortz M, Klimpke P, Kommer A, Grunder P, Steenken L, Dresel C, Kraus D, Schmidtmann I, Weinmann A, Weinmann-Menke J. Immunoadsorption study Mainz in adults with post-COVID syndrome (IAMPOCO)-a single-blinded sham-controlled crossover trial to evaluate the effect of immunoadsorption on post-COVID syndrome. Trials. 2025 Apr 3;26(1):119. doi: 10.1186/s13063-025-08825-7. PMID 40176165